CLINICAL TRIAL: NCT01335022
Title: African American Community Health Project on Cardiovascular Disease (AACP-CVD)
Brief Title: African American Community Health Project on Cardiovascular Disease
Acronym: AACP-CVD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Donald Lloyd-Jones, MD, ScM, FACC, FAHA, Northwestern University Department of Preventive Medicine & Cardiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU00035483
Record Dates: First submitted 2011-04-04; First posted 2011-04-13 (Estimated); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular Disease Education (Experimental): 6 lectures on cardiovascular disease were given over a 2 month time period
  Interventions: Behavioral: lecture

INTERVENTIONS:
Behavioral: lecture — 6 lectures on cardiovascular disease covering obesity, diet & exercise, smoking cessation, coronary artery disease, hypertension, heart failure, diabetes, peripheral vascular disease, and stroke.

SUMMARY:
The investigators seek to demonstrate that interactive physician-led education through partnership with an African American church will improve awareness and knowledge of cardiovascular disease in the African American community and will result in objective improvement in major risk factors associated with cardiovascular disease (CVD).

DETAILED DESCRIPTION:
Cardiovascular disease causes significant morbidity and mortality in the African American community. Among African Americans adults almost 1/3 have hypertension, 1/10 have heart disease, 1/20 have coronary heart disease, and 1/30 have had a stroke. Compared to their Caucasian American counterparts, African Americans are 3 times more times as likely to die from cardiovascular diseases than Caucasians, 1.5 times more likely to die from heart failure, and 1.8 times more likely to die from stroke. In addition, both lower socioeconomic position and minority race/ethnicity are associated with poorer health and shortened survival. These alarming statistics highlight the health disparities in the African American community. In our study, the investigators propose that interactive physician-led education through partnership with an African American church will improve awareness and knowledge of CVD in the African American community and will result in objective improvement in major risk factors associated with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* African American adults > 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 2 months
  Change after educational series
Weight | 2 months
  Change after educational series
Body mass index | 2 months
  Change after educational series
Waist Circumference | 2 months
  Change after educational series
Multiple choice test on cardiovascular disease | 2 months
  The multiple choice test is a 25-question test on general cardiovascular disease knowledge. It covers diet, exercise, smoking, obesity, coronary artery disease, heart failure, diabetes, stroke, and peripheral artery disease. This test is given at the start of the study and after the educational intervention. The overall test scores are compared by percentage correct. The individual questions are examined for group knowledge level on a particular topic. For example, the % correct of the group on a question about diabetes would reflect knowledge of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Lloyd-Jones, MD, ScM, Principal Investigator — Northwestern University; William J Mosley II, MD, Study Director — Northwestern University
Locations (1):
- Heritage International Christian Church, Chicago, Illinois, United States

REFERENCES:
- See also: Study Website — https://sites.google.com/site/drwilliamjmosleyii/